CLINICAL TRIAL: NCT01084109
Title: Complementary Feeding - A Global Network Cluster Randomized Controlled Trial
Brief Title: First Bites: Complementary Feeding - A Global Network Cluster Randomized Controlled Trial
Acronym: First Bites
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NICHD Global Network for Women's and Children's Health (Network)
Collaborators: Kinshasa School of Public Health (Other); University of Zambia (Other); INCAP, Chiimaltenango, Guatemala (Unknown); Aga Khan University (Other); University of Colorado, Denver (Other); University of North Carolina, Chapel Hill (Other); University of Alabama at Birmingham (Other); Drexel University (Other); RTI International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: GN CF
Record Dates: First submitted 2010-03-09; First posted 2010-03-10 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Complementary Feeding; Infant Growth
Keywords: Complementary feeding; Infant growth; Developing countries
MeSH Terms: interventions — Edible Grain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Daily intake of one half ounce of lyophilized meat between 6-18 months of age (0.5 oz for 6-12 mo; 0.75 oz for 12-18 mo)
  Interventions: Other: Lyophilized meat
- 2 (Active Comparator): Daily intake of an equi-caloric fortified cereal as complementary feed from 6 to 18 months.
  Interventions: Other: Cereal

INTERVENTIONS:
Other: Lyophilized meat — Daily intake of one half ounce of lyophilized meat between 6-18 months of age (0.5 oz for 6-12 mo; 0.75 oz for 12-18 mo)
  Arms: 1
Other: Cereal — Daily intake of an equi-caloric fortified cereal as complementary feed from 6 to 18 months.
  Arms: 2

SUMMARY:
The specific aims of this project is to determine the impact of a daily intake of one half ounce of lyophilized meat between 6-18 months of age (0.5 oz for 6-12 mo; 0.75 oz for 12-18 mo) on linear growth velocity, zinc and iron intakes and status, brain growth and neurocognitive development, and infectious disease morbidity in populations traditionally dependent on non-micronutrient fortified plant foods for complementary feeding.

DETAILED DESCRIPTION:
Inadequate and inappropriate complementary feeding are major factors contributing to excess morbidity and mortality in young children. Prominent among nutrient inadequacies are those of iron and zinc. While huge campaigns are being mounted to fortify complementary foods and to distribute supplements, the effectiveness of these programs is generally uncertain and they do not reach millions of rural poor. By comparison, little support is being given to local food-based solutions. These not only require diversity of plant foods but appear to require the inclusion of meat to achieve zinc and iron requirements. Local supplies of meat are achievable but only with a concerted international and local effort. To justify this effort requires a multi-site efficacy study, the results of which, if positive, will leave no doubt that the effort required to provide sustainable local sources of meat for complementary feeds is worthwhile. The principal hypothesis to be tested is that daily intake of beef (1 oz/d for 6-12 mo and 1.5 oz/d for 12-18 mo) added to usual primarily plant-derived complementary feeds plus selected repetitive nutrition education messages results in greater linear growth velocity than does a micronutrient (including Zn and Fe) fortified equi-caloric cereal/legume supplement plus the same educational messages. Participants from four sites in the Global Network which have stunting rates > 20%, i.e. Guatemala, Pakistan and Zambia will be randomized by clusters to receive either ½ oz lyophilized beef (equivalent to 1 oz cooked beef)/d or the equi-caloric micronutrient-fortified plant-based supplement (both increasing by 50% at age 1 year). Both groups will receive three repetitive messages delivered by study coordinators and through the local health system as part of integrated health care. These are: provide a thick puree/gruel; feed complementary foods at least three times per day; and maximize dietary diversity. These interventions will be preceded by messages to promote exclusive breast feeding until 6 months and to start complementary feeding promptly at that time as far as possible. The meat or fortified cereal supplement will be provided daily in a group setting for each cluster; as necessary the food intervention and messages will be delivered at home by the assigned community coordinator or alternate. Outcome measures, obtained by a separate group of local, trained assessment workers, include: longitudinal linear growth between 6-18 months (primary outcome); weight and head circumference; assessment of dietary variety and diversity at 6,9,12, and 18 months; indices of iron, zinc and Vitamin B12 status at 18 months; neurocognitive development at 18 months; and incidence of diarrhea and lower respiratory infections. A positive multi-country, multi-culture outcome of this trial will demonstrate the efficacy of a regular intake of meat commencing at age 6 months to achieve nutritionally complete complementary feeding and will provide a strong rationale for global efforts to enhance local supplies of meat and achieve acceptance of meats as complementary food.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for clusters: Each cluster will be a rural community characterized by inhabitants with low income and served by one community health center. A primary criterion is that national or other available statistics indicate a prevalence of stunting (mean length for age Z-scores in second year < -2) of at least 20% in young children.
* Inclusion criteria for individual families:

  * Infant aged 3-4 months;
  * Primarily or exclusively breast feeding with intent to continue breast feeding through at least 1 year.

Exclusion Criteria:

* Exclusion criteria for individual families: Exclusion criteria include any population/family that is receiving or likely to receive free or subsidized complementary foods (or infant formula) through the health system or NGOs; any individual families who are feeding or intend to feed fortified infant formula or micronutrient-fortified commercial complementary foods.
* Exclusion criteria for infants: Infants meeting the following criteria will be excluded from participation:

  1. known congenital anomaly;
  2. infant of multiple births;
  3. known neurological deficit apparent at the time of enrollment (including seizures).

Ages: 3 Months to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1236 (Actual)
Dates: Start 2008-07; Primary Completion 2010-04 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Linear growth velocity | 6 to 18 months of age

SECONDARY OUTCOMES:
Infant Zinc and Ferritin levels | 18 months
Bayleys II | 18 months
Incidence of diarrhea, lower respiratory infection, and malaria | 6 to 18 months

CONTACTS AND LOCATIONS:
Locations (4):
- Institute for Nutrition of Central America and Panama (INCAP), Chiimaltenango, Guatemala
- Agha Khan University, Karachi, Pakistan
- Kinshasa School of Public Health, Karawa, Republic of the Congo
- University of Zambia, Lusaka, Zambia

REFERENCES:
- [Derived] Manasyan A, Salas AA, Nolen T, Chomba E, Mazariegos M, Tshefu Kitoto A, Saleem S, Naqvi F, Hambidge KM, Goco N, McClure EM, Wallander JL, Biasini FJ, Goldenberg RL, Bose CL, Koso-Thomas M, Krebs NF, Carlo WA. Diagnostic accuracy of ASQ for screening of neurodevelopmental delays in low resource countries. BMJ Open. 2023 May 23;13(5):e065076. doi: 10.1136/bmjopen-2022-065076. PMID 37221030
- [Derived] Krebs NF, Mazariegos M, Chomba E, Sami N, Pasha O, Tshefu A, Carlo WA, Goldenberg RL, Bose CL, Wright LL, Koso-Thomas M, Goco N, Kindem M, McClure EM, Westcott J, Garces A, Lokangaka A, Manasyan A, Imenda E, Hartwell TD, Hambidge KM. Randomized controlled trial of meat compared with multimicronutrient-fortified cereal in infants and toddlers with high stunting rates in diverse settings. Am J Clin Nutr. 2012 Oct;96(4):840-7. doi: 10.3945/ajcn.112.041962. Epub 2012 Sep 5. PMID 22952176
- [Derived] Krebs NF, Hambidge KM, Mazariegos M, Westcott J, Goco N, Wright LL, Koso-Thomas M, Tshefu A, Bose C, Pasha O, Goldenberg R, Chomba E, Carlo W, Kindem M, Das A, Hartwell T, McClure E; Complementary Feeding Study Group. Complementary feeding: a Global Network cluster randomized controlled trial. BMC Pediatr. 2011 Jan 13;11:4. doi: 10.1186/1471-2431-11-4. PMID 21232139